CLINICAL TRIAL: NCT04084197
Title: An Open-label, Randomized, Single-dose Crossover Study to Evaluate the Pharmacokinetics, Safety and Tolerability of HIP1801 in Healthy Male Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety and Tolerability of HIP1801 in Healthy Male Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-TOD-101
Record Dates: First submitted 2019-09-09; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Experimental): Period 1 : Fasted state + HIP1402, Period 2 : Fasted state + HIP1801
  Interventions: Drug: HIP1402; Drug: HIP1801
- Sequence 2 (Experimental): Period 1 : Fasted state + HIP1801, Period 2 : Fasted state + HIP1402
  Interventions: Drug: HIP1402; Drug: HIP1801
- Sequence 3 (Experimental): High fat diet + HIP1402, Period 2 : High fat diet + HIP1801
  Interventions: Drug: HIP1402; Drug: HIP1801
- Sequence 4 (Experimental): High fat diet + HIP1801, Period 2 : High fat diet + HIP1402
  Interventions: Drug: HIP1402; Drug: HIP1801

INTERVENTIONS:
Drug: HIP1402 — Tamsulosin (HanmiTams Capsule) 0.4mg
Drug: HIP1801 — Tamsulosin 0.4mg

SUMMARY:
An open-label, randomized, single-dose crossover study to evaluate the pharmacokinetics, safety and tolerability of HIP1801 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19~45 years in healthy male volunteers
2. BMI is more than 18.5 kg/m^2 , no more than 29.9 kg/m^2
3. Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
2. Subjects who judged ineligible by the investigator

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 1.Age 19~45 years in healthy male volunteers
Enrollment: 61 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-04 (Actual)

PRIMARY OUTCOMES:
Cmax of Tamsulosin | pre-dose(0 hour), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
AUClast of Tamsulosin | pre-dose(0 hour), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation

SECONDARY OUTCOMES:
AUCinf of Tamsulosin | pre-dose(0 hour), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
Tmax of Tamsulosin | pre-dose(0 hour), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
t1/2 of Tamsulosin | pre-dose(0 hour), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
CL/F of Tamsulosin | pre-dose(0 hour), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
Vd/F of Tamsulosin | pre-dose(0 hour), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No